CLINICAL TRIAL: NCT00476593
Title: Retinal Optical Coherence Tomography and Multifocal Electroretinogram; Establishing Normal Ranges Related to Age and Reproductive Factors; With the Use of Anti-inflammatory Medications;In Uncomplicated Anterior Uveitis; Anatomy and Function.
Brief Title: Retinal OCT and (mfERG) Related to Age, Sex, and the Use of Anti-inflammatory Medications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 47026200; NSD 200500943 (Other: Helse Midt-Norge); REK 4.2005.13 (Other: Helse Midt-Norge)
Record Dates: First submitted 2007-05-21; First posted 2007-05-22 (Estimated); Results first posted 2011-06-22 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2017-03

CONDITIONS: Uveitis; Iritis; Iridocyclitis; Anterior Uveitis; Macular Edema
Keywords: Uveitis; Iritis; Macular Thickness; HLA-B27 related; Macular edema; Macular thickening; OCT; mfERG; Eye drops; Dexamethosone; Diclofenac; Retinal aging
MeSH Terms: conditions — Uveitis; Iritis; Iridocyclitis; Uveitis, Anterior; Macular Edema | interventions — Diclofenac; Ophthalmic Solutions; Dexamethasone; dexamethasone 21-phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diclofenac (Experimental): Preservative- free Diclofenac Na 0.1 % eye drops were applied in one consecutively assigned eye of healthy volunteers four times a day for three days, after which macular thichness was measured in both subjects' eyes with the OCT .
  Interventions: Drug: Diclofenac
- Dexamethasone (Experimental): Benzalkonium-reserved Dexamethasone Sodium Phosphate 0.1% was applied in one consecutively assigned eye of healthy volunteers six times a day for three days, after which macular thickness was assessed in both subjects's eyes with the OCT.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Diclofenac — Preservative- free Diclofenac Na 0.1% eye drops (Voltaren Ophta SDU;Novartis Pharms). One drop four times daily in one eys for three days.
  The evaluation of macular thickness/function after 3 days use of anti-inflammatory eye drops in healthy subjects is the only sub-study involving an intervention design.
  Other Names: Voltaren (Ophta SDU;Novartis Pharms) eye drops.
  Arms: Diclofenac
Drug: Dexamethasone — Dexamethasone sodium phosphate 0.1% eye drops (Spersadex OmniVision, Novartis Pharma), one drop six times daily for three days in one eye.
  Pharms). One drop four times daily in one eys for three days.
  The evaluation of macular thickness/function after 3 days use of anti-inflammatory eye drops in healthy subjects is the only sub-study involving an intervention design.
  Other Names: Spersadex (OmniVision, Novartis Pharma)eye drops.
  Arms: Dexamethasone

SUMMARY:
Retinal optical coherence tomography (OCT) is an established technology which enables a detailed cross-sectional visualization of the retinal micro-anatomy, and an objective measurement of its thickness in-vivo. Multifocal electroretinogram (MfERG) measures function of the central retina. Both technologies are relatively new and they provide complimentary to each other information on retinal anatomy and function.

The aims of this study is to establish normal ranges for OCT and mfERG measurements related to age, gender and reproductive factors such as parity and the use of contraception in Norwegians; to assess the presumably healthy central retina with the use of anti-inflammatory medication with relation to age and sex ; to study the frequency and extent of retinal thickening and change in retinal function in patients with anterior uveitis not complicated with macular edema; to assess whether the presence of the HLA-B27 haplotype or uveitis recidive affects macular thickening/function in uveitis.

DETAILED DESCRIPTION:
Normal optical coherence tomography (OCT) and Multifocal electroretinogram (MfERG) measurements may vary with race, age, sex, parity and the use of hormone therapy in health. It has therefore been recommended to gather normative data on the individual OCT/MfERG equipment in each laboratory. This is the reason why we gathered our local normative material on both machines. We also assessed our normative material on the OCT in relation to age, sex, parity and the use of contraception for future matching with patients.

It has been hypothesized that para-inflammation states are involved in retinal aging in health. We assume that the age-related changes we observed in our normative OCT material are related to low-grade chronic inflammation in the retina. We therefore assessed the effect of to commercially available anti-inflammatory eye drops- diclofenac and dexamethasone,which are often used in inflammation-related states in ophthalmology for their effect on macular thickness in health and with aging.

Uveitis is a frank intraocular inflammation which may lead to macular edema. Macular edema is often transient in uveitis and its presence has been previously reported in severe or long-lasting uveitis. In some cases mecular edema may become chronic or refractory to treatment. However, whether uncomplicated anterior uveitis with no clinically evident macular edema leads to macular thickening detectable with the OCT, or whether monolateral uveitis may cause bilateral macular thickening is not known. We therefore assesed both eyes of patients with anterior uveitis for macular thickening with the OCT.

To correlate macular anatomy with its function some subjects included in the OCT study were also examined with the mfERG. However, at present the MfERG result have not been analyzed.

ELIGIBILITY:
Inclusion Criteria:

Adults healthy volunteers and adult patients with anterior uveitis who wish to participate.

Exclusion Criteria:

* Patients with anterior uveitis who have other systemic diseases/conditions not related to their anterior uveitis, like high blood pressure, diabetes or epilepsy.
* Patients with ocular comorbidity or compliactions to their anterior uveitis, such as elevated ocular pressure or glaucoma.
* Previous or current macular edema or other posterior segment complications related to uveitis.
* Subjects with visual acuity worse than 0.8
* Subjects/patients with cataracts or other ocular media opacities
* Subjects/patients who are allergic to local anesthesia or mydriatics.
* Subjects/patients with high myopia/hyperopia
* Subjects/patients who have had intraocular surgery, although previous uncomplicated LASIK correction for low-grade myopia were accepted.
* Subjects/patients who cooperate poorly.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2005-09 (Actual); Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tor B Elsås, Professor, Study Director — Department of Ophthalmology, St. Olavs University Hospital, Trondheim, Norway; Trond Sand, Professor, Study Chair — Department of Neuroscience, Norwegian University of Science and Technology, Trondheim, Norway; Alexandra Wexler, Dr, Principal Investigator — Department of Neuroscience, Norwegian University of Science and Technology, Trondheim, Norway
Locations (2):
- Norway (2):
  - Department of Ophthalmology, St Olavs University Hospital, Trondheim
  - Department of Neuroscience, Norwegian University of Science and Technology, Trondheim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wexler A, Sand T, Elsas TB. Macular thickness measurements in healthy Norwegian volunteers: an optical coherence tomography study. BMC Ophthalmol. 2010 May 13;10:13. doi: 10.1186/1471-2415-10-13. PMID 20465801

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy subjects were recruited from students and staff at St. Olavs University Hospital and NTU for ophthalmic examination at the Department of Ophthalmology and mfERG testing at NTU, May 05- Sept. 07. From Sept.07 -sept.08 patients with uveitis were recruited from the Dep. of Opthalmology, healthy volunteers- both for OCT examination at the Dep.
Pre-assignment Details: We chose to focus primary on the OCT results because mfERG equipement was moved and its software was updated. MfERG results will be analyzed later. The main reason for participant exclusion in this study was either bad OCT scan quality or participant withdrawal because examinations turned out to be more time consuming then they thought.
Groups:
- A Diclofenac: Preservative- free Diclofenac Na 0.1 % eye drops were applied in one consecutively assigned eye of healthy volunteers four times a day for three days, after which macular thichness was measured in both subjects' eyes with the OCT .
- B Dexamethasone: Benzalkonium-reserved Dexamethasone Sodium Phosphate 0.1% was applied in one consecutively assigned eye of healthy volunteers six times a day for three days, after which macular thickness was assessed in both subjects's eyes with the OCT.
- Patients With Anterior Uveitis: Patients with anterior uveitis were recruited from the Department of Ophthalmology. They were treated for their uveitis and OCT scans of their both eyes were taken on follow up.
- Healthy Volunteers: Healthy volunteers recruited from students and staff at St Olavs University hospital and NTU went through an opthalmologic examination and OCT scans were taken of their both eyes. This groups was to serve as healthy controls and as matching normative data for patients
Period: Overall Study
Arm/Group | A Diclofenac | B Dexamethasone | Patients With Anterior Uveitis | Healthy Volunteers
Started | 32 | 19 | 38 | 129
Completed | 22 (all subjects completed treatment in one eye. However, bilateral OCT scans included only in 22 cases) | 17 (all subjects completed treatment in one eye. However, bilateral OCT scans included only in 17 cases) | 30 | 107
Not Completed | 10 | 2 | 8 | 22
Not completed — Lost to Follow-up | 10 | 2 | 8 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A Diclofenac | B Dexamethasone | Patients With Anterior Uveitis | Healthy Volunteers | Total
Number analyzed (Participants) | 22 | 17 | 30 | 107 | 176
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 22 | 17 | 29 | 107 | 175
  >=65 years | 0 | 0 | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.2 (10.9) | 46.2 (11.4) | 40.5 (2.3) | 42.4 (11.8) | 45.1 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 15 | 62 | 105
  Male | 7 | 4 | 15 | 45 | 71
Region of Enrollment [Number; unit: participants]
  Norway | 22 | 17 | 30 | 107 | 176

OUTCOME MEASURES:

1. Primary Outcome: Macular Thickness Measured With the OCT; in Relation to Age, Sex, Reproductive Factors and the Use of Anti-inflammatory Eye Drops in Health; in Uncomplicated Anterior Uveitis.
Description: Macular thickness was assessed with the OCT in healthy subjects and in patients with anterior uveitis. Data was analyzed with respect to age, sex, parity, the use of hormonal therapy, after treatment with to types of anti-inflammatory eye drops, and in uncomplicated uveitis.
Time Frame: Macular thickness measured with the OCT
Population: Enrolled healthy subjects and patients with anterior uveitis who volunteered through enrollment period
Measure: Mean (Standard Deviation); unit: Macular Thickness in micron
Arm/Group | A Diclofenac | B Dexamethasone | Patients With Anterior Uveitis | Healthy Volunteers
Number analyzed (Participants) | 22 | 17 | 30 | 107
Macular Thickness in micron | 268 (13) | 272 (16) | 276 (21) | 267 (13)
Statistical Analysis 1: Comparison: A Diclofenac vs B Dexamethasone; Subjects who received diclofenac or dexamethasone eye drops in one eye. Macular thickness in both were compared between same subjects' eyes after 3 day's treatment. Diclofenac and dexamethasone treated eyes were not compared with each other, but with the contralateral eye of same subject by a paired Student's t-test in each medication group; Test type: Superiority or Other; p = 0.018, t-test, 2 sided — Hypothesis: the use of diclofenac/dexamethasone does not influence macular thickness in treated eyes compared with untreated eyes of same subject; The possible effect of both anti-inflammatory medications was tested in relation to participants' age and gender
Statistical Analysis 2: Comparison: Patients With Anterior Uveitis vs Healthy Volunteers; Patient's healthy eyes were compared with sex and age matched healthy controls with Two Sample Student't t-test. Null hypothesis was that quiet, currently unaffected eyes of patients had same macular thickness as age and sex matched controls; Test type: Superiority or Other; p = 0.024, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | A Diclofenac | B Dexamethasone | Patients With Anterior Uveitis | Healthy Volunteers
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes